CLINICAL TRIAL: NCT06798662
Title: Multimodal Nerve Block and Pulse Radiofrequency for Acute Herpes Zoster Pain: a Prospective, Randomized, Controlled, Triple-blind Trial
Brief Title: Multimodal Nerve Block and Pulse Radiofrequency for Acute Herpes Zoster Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaguang Duan (Other)
Responsible Party: Sponsor-Investigator, Xiaguang Duan, Deputy Chief of Anesthesiology, Inner Mongolia Baogang Hospital
Organization: Inner Mongolia Baogang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-MER-314
Record Dates: First submitted 2025-01-17; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Herpes Zoster (HZ)
MeSH Terms: conditions — Herpes Zoster | interventions — Dental Occlusion; Pharmaceutical Preparations; Famciclovir; Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- RISS group (Experimental): Rhomboid Intercostal and Subserratus Plane (RISS) Block:
  The RISS block is a composite nerve block technique that involves two injection sites: the inter-rhomboid plane and the sub-serratus plane. The selection of block plane was determined by the patient's specific location of pain.
  Rhomboid Intercostal Plane Block (RIPB):
  For the Rhomboid Intercostal Plane Block (RIPB), a high-frequency linear ultrasound transducer was initially positioned in a sagittal orientation, medial to the scapular border. It was then slightly rotated to obtain an oblique sagittal view (oblique paramedian sagittal view), located 1-2 cm lateral to the scapular border. Upon obtaining the appropriate ultrasound image, the following anatomical structures were identified sequentially, from superficial to deep: the trapezius muscle, the rhomboid muscles (specifically, the major rhomboid), the intercostal muscles (located between the ribs), the pleura, and the lung. The target injection plane was the fascial plan
  Interventions: Device: Rhomboid Intercostal and Subserratus Plane (RISS) Block (2% ropivacaine or 133 mg of liposomal bupivacaine); Drug: Drug (famciclovir and gabapentin)
- PVB group (Experimental): For the Paravertebral (PVB) block, a high-frequency linear ultrasound transducer was placed transversely, parallel to the spinous processes, approximately 2-3 cm lateral to the spinous process of the target thoracic vertebral segment. The position and angle of the transducer were adjusted to clearly visualize the transverse process (TP) and the axial view of the lamina of the target vertebra. In the ultrasound image, the transverse process appeared as a hyperechoic structure, typically with a characteristic acoustic shadow posterior to it. Subsequently, the transducer was slightly slid caudally, causing the transverse process and its acoustic shadow to gradually disappear from view. At this point, the ultrasound image revealed components of the paravertebral space (PVS), including the parietal pleura, the superior costotransverse ligament, and the intercostal fascia, which exhibited a heterogeneous mixed echogenicity. Using an in-plane technique, a puncture needle was advanced from la
  Interventions: Device: Paravertebral (PVB) Block (2% ropivacaine or 133 mg of liposomal bupivacaine); Drug: Drug (famciclovir and gabapentin)
- ICN group (Experimental): The patient is positioned in either the lateral decubitus or sitting position, with the affected side facing upwards, ensuring adequate exposure of the targeted intercostal region. A high-frequency linear ultrasound transducer is placed transversely over the posterior lateral aspect of the targeted rib, using the vertebral column as a reference point. The transducer is then scanned laterally to identify the target rib, clearly visualizing the rib, intercostal muscles, and pleura. The intercostal nerve appears as a small hyperechoic structure located between the internal and innermost intercostal muscles. The needle is advanced until it contacts the inferior border of the rib. The needle is then slightly withdrawn and positioned between the internal and innermost intercostal muscles to avoid pleural puncture. After negative aspiration, 10 mL of 0.5% ropivacaine (or 133 mg of liposomal bupivacaine) combined with 10 mg of triamcinolone acetonide is injected slowly.
  Interventions: Device: Intercostal nerve block (2% ropivacaine or 133 mg of liposomal bupivacaine); Drug: Drug (famciclovir and gabapentin)
- PRF group (Experimental): A high-frequency linear ultrasound transducer will be used for this procedure. The transducer will be placed transversely over the target rib area to obtain a clear visualization of the rib, intercostal muscles, and pleura. The entry point for needle insertion will be selected 1-2 cm inferior to the inferior border of the target rib. Using a 22G radiofrequency (RF) needle, an in-plane approach will be used for needle advancement. The needle will be advanced slowly until it reaches the inferior border of the rib. The needle will then be withdrawn 1-2 mm to ensure the needle tip is positioned adjacent to the intercostal nerve. The RF needle will then be connected to the RF generator for sensory testing. Stimulation parameters will be set at 50 Hz and 0.5-1V. The target location will be considered accurate if stimulation induces pain in the participant. Pulsed radiofrequency treatment will then be administered using the following parameters: voltage of 45V, frequency of 2 Hz, pulse width
  Interventions: Device: Ultrasound-Guided Pulsed Radiofrequency (PRF); Drug: Drug (famciclovir and gabapentin)

INTERVENTIONS:
Device: Ultrasound-Guided Pulsed Radiofrequency (PRF) — A high-frequency linear ultrasound transducer will be used for this procedure. The transducer will be placed transversely over the target rib area to obtain a clear visualization of the rib, intercostal muscles, and pleura. The entry point for needle insertion will be selected 1-2 cm inferior to the inferior border of the target rib. Using a 22G radiofrequency (RF) needle, an in-plane approach will be used for needle advancement. The needle will be advanced slowly until it reaches the inferior border of the rib. The needle will then be withdrawn 1-2 mm to ensure the needle tip is positioned adjacent to the intercostal nerve. The RF needle will then be connected to the RF generator for sensory testing. Stimulation parameters will be set at 50 Hz and 0.5-1V. The target location will be considered accurate if stimulation induces pain in the participant. Pulsed radiofrequency treatment will then be administered using the following parameters: voltage of 45V, frequency of 2 Hz, pulse width
  Arms: PRF group
Device: Intercostal nerve block (2% ropivacaine or 133 mg of liposomal bupivacaine) — The patient is positioned in either the lateral decubitus or sitting position, with the affected side facing upwards, ensuring adequate exposure of the targeted intercostal region. A high-frequency linear ultrasound transducer is placed transversely over the posterior lateral aspect of the targeted rib, using the vertebral column as a reference point. The transducer is then scanned laterally to identify the target rib, clearly visualizing the rib, intercostal muscles, and pleura. The intercostal nerve appears as a small hyperechoic structure located between the internal and innermost intercostal muscles. The needle is advanced until it contacts the inferior border of the rib. The needle is then slightly withdrawn and positioned between the internal and innermost intercostal muscles to avoid pleural puncture. After negative aspiration, 10 mL of 0.5% ropivacaine (or 133 mg of liposomal bupivacaine) combined with 10 mg of triamcinolone acetonide is injected slowly.
  Arms: ICN group
Device: Paravertebral (PVB) Block (2% ropivacaine or 133 mg of liposomal bupivacaine) — For the Paravertebral (PVB) block, a high-frequency linear ultrasound transducer was placed transversely, parallel to the spinous processes, approximately 2-3 cm lateral to the spinous process of the target thoracic vertebral segment. The position and angle of the transducer were adjusted to clearly visualize the transverse process (TP) and the axial view of the lamina of the target vertebra. In the ultrasound image, the transverse process appeared as a hyperechoic structure, typically with a characteristic acoustic shadow posterior to it. Subsequently, the transducer was slightly slid caudally, causing the transverse process and its acoustic shadow to gradually disappear from view. At this point, the ultrasound image revealed components of the paravertebral space (PVS), including the parietal pleura, the superior costotransverse ligament, and the intercostal fascia, which exhibited a heterogeneous mixed echogenicity. Using an in-plane technique, a puncture needle was advanced from lat
  Arms: PVB group
Device: Rhomboid Intercostal and Subserratus Plane (RISS) Block (2% ropivacaine or 133 mg of liposomal bupivacaine) — The RISS block is a composite nerve block technique that involves two injection sites: the inter-rhomboid plane and the sub-serratus plane. The selection of block plane was determined by the patient's specific location of pain.
  Rhomboid Intercostal Plane Block (RIPB):
  For the Rhomboid Intercostal Plane Block (RIPB), a high-frequency linear ultrasound transducer was initially positioned in a sagittal orientation, medial to the scapular border. It was then slightly rotated to obtain an oblique sagittal view (oblique paramedian sagittal view), located 1-2 cm lateral to the scapular border. Upon obtaining the appropriate ultrasound image, the following anatomical structures were identified sequentially, from superficial to deep: the trapezius muscle, the rhomboid muscles (specifically, the major rhomboid), the intercostal muscles (located between the ribs), the pleura, and the lung. The target injection plane was the fascial plane situated between the rhomboid muscle and the intercostal
  Arms: RISS group
Drug: Drug (famciclovir and gabapentin) — All patients will receive famciclovir and gabapentin. All participants will receive standard antiviral therapy with famciclovir 500 mg orally three times daily for 7 days. Gabapentin will be initiated at a typical starting dose of 300 mg per day, administered in three divided doses. The dosage may be gradually increased, as needed and tolerated, up to a maximum dose of 1800 mg per day.

SUMMARY:
The primary objective of this clinical trial is to evaluate the efficacy of liposomal bupivacaine and ropivacaine in the treatment of pain associated with herpes zoster (shingles). This trial will also assess the safety profiles of both liposomal bupivacaine and ropivacaine.

The study aims to address the following key questions:

Does nerve blockade with liposomal bupivacaine or ropivacaine reduce the required dosage of gabapentin in participants? What medical issues, if any, arise in participants undergoing paravertebral block, intercostal nerve block, RISS (Radiofrequency Intervention for Spinal Segment); or pulsed radiofrequency (PRF)? Can nerve blocks, specifically paravertebral block, intercostal nerve block, RISS; and PRF, effectively treat severe postherpetic neuralgia (PHN)? The study will compare these interventions.

Study Procedures:

Participants will:Receive ultrasound-guided nerve blocks or pulsed radiofrequency every 48 hours, for a total of 3 treatments.

Undergo assessments, either in-person or via telephone, at the following time points: before therapy (baseline), on the day of treatment (Day 1), Day 7, Day 30, and Day 90 post-treatment.

Have their symptoms recorded, along with their scores on the Numerical Rating Scale (NRS) and the Zoster Brief Pain Inventory (ZBPI).

DETAILED DESCRIPTION:
Study design：This study is a prospective, randomized, controlled, comparative trial with blinding of both participants and clinicians. The trial is designed to assess both the superiority and non-inferiority of several interventions for analgesia in postherpetic neuralgia (PHN). The following interventions will be compared: Rhomboid Intercostal and Subserratus Plane (RISS) block, Paravertebral (PVB) block, Intercostal nerve block, Pulsed radiofrequency (PRF). Participant recruitment will take place at Baogang Hospital in Inner Mongolia. This study has been approved by the Medical Ethics Committee of Baogang Hospital, Inner Mongolia. The research will be conducted in accordance with the principles outlined in the Declaration of Helsinki and the Consolidated Standards of Reporting Trials (CONSORT) guidelines. All participants will provide voluntary, informed consent prior to enrollment.

Patients：A total of 120 patients, aged 44 to 82 years, with an American Society of Anesthesiologists (ASA) physical status classification of I-III, who are scheduled to receive treatment for pain associated with herpes zoster (shingles) with either Rhomboid Intercostal and Subserratus Plane (RISS) block, Paravertebral (PVB) block, intercostal nerve block, or pulsed radiofrequency (PRF), will be enrolled in the study between February 2025 and May 2025. Patients will be randomly assigned to one of four groups, with 30 patients in each group.

Randomization and Blinding：This study employed block randomization to generate the random allocation sequence. A block size of 6 was set, and the random sequence was generated using dedicated software (the blockrand package in R version 4.3.2). The allocation of the random sequence was performed by an independent third party, and allocation concealment was implemented using sequentially numbered, sealed, opaque envelopes. The research team remained blinded throughout the randomization process and was not involved in the generation or allocation of the random sequence.

Intervention：For patients with postherpetic neuralgia (PHN) unresponsive to pharmacotherapy, consideration will be given to the Rhomboid Intercostal and Subserratus Plane (RISS) block, Paravertebral (PVB) block, intercostal nerve block, or pulsed radiofrequency (PRF). All patients will receive famciclovir and gabapentin. All participants will receive standard antiviral therapy with famciclovir 500 mg orally three times daily for 7 days. Gabapentin will be initiated at a typical starting dose of 300 mg per day, administered in three divided doses. The dosage may be gradually increased, as needed and tolerated, up to a maximum dose of 1800 mg per day. All procedures will be performed in an outpatient surgical suite. All participating physicians will have undergone standardized training. Upon entering the procedure room, patients will have electrocardiogram (ECG), blood pressure, and oxygen saturation monitoring established. Patients will be positioned in the prone position with their arms abducted and internally rotated. Ultrasound guidance will be utilized with a SonoSite Edge II ultrasound system (Fujifilm SonoSite, Bothell, WA, USA) equipped with a linear 13-6 MHz transducer (HFL50x; Fujifilm SonoSite, Bothell, WA, USA). For each nerve block, a 5 mL test dose will be administered initially, and clinical signs of pain relief in the affected thoracic dermatome will be observed. After confirmation of appropriate injection site, the remaining medication will be administered. Patients will receive ultrasound-guided nerve blocks every 48 hours for a total of 3 treatments.

Rhomboid Intercostal and Subserratus Plane (RISS) Block:

The RISS block is a composite nerve block technique that involves two injection sites: the inter-rhomboid plane and the sub-serratus plane. The selection of block plane was determined by the patient's specific location of pain.

Rhomboid Intercostal Plane Block (RIPB):

For the Rhomboid Intercostal Plane Block (RIPB), a high-frequency linear ultrasound transducer was initially positioned in a sagittal orientation, medial to the scapular border. It was then slightly rotated to obtain an oblique sagittal view (oblique paramedian sagittal view), located 1-2 cm lateral to the scapular border. Upon obtaining the appropriate ultrasound image, the following anatomical structures were identified sequentially, from superficial to deep: the trapezius muscle, the rhomboid muscles (specifically, the major rhomboid), the intercostal muscles (located between the ribs), the pleura, and the lung. The target injection plane was the fascial plane situated between the rhomboid muscle and the intercostal muscle. Following confirmation of correct needle tip placement, a solution of 10 mL of 0.5% ropivacaine (or 133 mg of liposomal bupivacaine) combined with 10 mg of triamcinolone acetonide was slowly injected in divided doses. The injection was performed under real-time ultrasound visualization, and the spread of the local anesthetic was carefully observed to ensure adequate distribution within the target fascial plane.

Subserratus Plane Block (SSPB):

For the Subserratus Plane Block (SSPB), the ultrasound transducer was moved inferiorly, to the caudal aspect of the inferior angle of the scapula, and then laterally, to a point posterior to the posterior axillary line. In the ultrasound image, the following structures were visualized sequentially, from superficial to deep: the latissimus dorsi muscle, the serratus anterior muscle, the intercostal muscles (located between the ribs), the pleura, and the lung. The target injection plane was the fascial plane between the serratus anterior muscle and the external intercostal muscle. Following confirmation of correct needle tip placement, a solution of 15 mL of 0.5% ropivacaine (or 133 mg of liposomal bupivacaine) combined with 10 mg of triamcinolone acetonide was slowly injected in divided doses. The injection was performed under real-time ultrasound visualization, and the spread of the local anesthetic was carefully observed to ensure adequate distribution within the target fascial plane and to cover the surface of the intercostal muscles.

Paravertebral (PVB) Block:

For the Paravertebral (PVB) block, a high-frequency linear ultrasound transducer was placed transversely, parallel to the spinous processes, approximately 2-3 cm lateral to the spinous process of the target thoracic vertebral segment. The position and angle of the transducer were adjusted to clearly visualize the transverse process (TP) and the axial view of the lamina of the target vertebra. In the ultrasound image, the transverse process appeared as a hyperechoic structure, typically with a characteristic acoustic shadow posterior to it. Subsequently, the transducer was slightly slid caudally, causing the transverse process and its acoustic shadow to gradually disappear from view. At this point, the ultrasound image revealed components of the paravertebral space (PVS), including the parietal pleura, the superior costotransverse ligament, and the intercostal fascia, which exhibited a heterogeneous mixed echogenicity. Using an in-plane technique, a puncture needle was advanced from lateral to medial under real-time ultrasound guidance towards the target paravertebral space. The needle was carefully advanced, passing through the intercostal fascia, while avoiding the parietal pleura, and positioning the needle tip superior to the costotransverse ligament. Following confirmation of correct needle tip placement, a solution of 10 mL of 0.5% ropivacaine (or 133 mg of liposomal bupivacaine) combined with 10 mg of triamcinolone acetonide was slowly injected in divided doses. The injection was performed under real-time ultrasound visualization, and the spread of the local anesthetic was carefully observed to ensure adequate distribution within the PVS for an effective block. If multiple nerves were involved, the injection sites were spaced one thoracic vertebral segment apart.

Intercostal Nerve Block:

The patient is positioned in either the lateral decubitus or sitting position, with the affected side facing upwards, ensuring adequate exposure of the targeted intercostal region. A high-frequency linear ultrasound transducer is placed transversely over the posterior lateral aspect of the targeted rib, using the vertebral column as a reference point. The transducer is then scanned laterally to identify the target rib, clearly visualizing the rib, intercostal muscles, and pleura. The intercostal nerve appears as a small hyperechoic structure located between the internal and innermost intercostal muscles. The needle is advanced until it contacts the inferior border of the rib. The needle is then slightly withdrawn and positioned between the internal and innermost intercostal muscles to avoid pleural puncture. After negative aspiration, 10 mL of 0.5% ropivacaine (or 133 mg of liposomal bupivacaine) combined with 10 mg of triamcinolone acetonide is injected slowly.

Ultrasound-Guided Pulsed Radiofrequency (PRF):

A high-frequency linear ultrasound transducer will be used for this procedure. The transducer will be placed transversely over the target rib area to obtain a clear visualization of the rib, intercostal muscles, and pleura. The entry point for needle insertion will be selected 1-2 cm inferior to the inferior border of the target rib. Using a 22G radiofrequency (RF) needle, an in-plane approach will be used for needle advancement. The needle will be advanced slowly until it reaches the inferior border of the rib. The needle will then be withdrawn 1-2 mm to ensure the needle tip is positioned adjacent to the intercostal nerve. The RF needle will then be connected to the RF generator for sensory testing. Stimulation parameters will be set at 50 Hz and 0.5-1V. The target location will be considered accurate if stimulation induces pain in the participant. Pulsed radiofrequency treatment will then be administered using the following parameters: voltage of 45V, frequency of 2 Hz, pulse width of 20 ms, and treatment time of 360 seconds.

Outcomes and measures：Follow-up assessments will be conducted at the pain clinic by two specially trained nurses who are blinded to participant treatment allocation. Assessments will be performed at the following time points: prior to therapy (baseline), on the day of treatment (Day 1), Day 7 post-treatment, Day 30 post-treatment, and Day 90 post-treatment. These assessments will be conducted either in-person or via telephone.

ELIGIBILITY:
Inclusion Criteria:

* Presence of typical clinical manifestations of herpes zoster (shingles), including vesicular and painful rash.
* Diagnosis of postherpetic neuralgia (PHN) lasting for more than one month, unresponsive to conventional treatment.
* Visual Analog Scale (VAS) score ≥ 4.
* Involvement of thoracic nerve roots.

Exclusion Criteria:

* Refusal to provide written informed consent.
* Inability to cooperate with study assessments.
* History of systemic autoimmune disease, organ transplantation, or cancer.
* Prior receipt of other invasive pain treatments, such as spinal cord stimulation.
* Presence of a central nervous system (CNS) disorder.
* Presence of coagulopathy.
* Skin infection at the puncture site.
* Pregnancy or breastfeeding.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-10 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale(NRS) | At baseline (before therapy), at 1 day of treatment, at 7 days post-treatment, 30 days post-treatment, and 90 days post-treatment
  The NRS, Numerical Rating Scale, is a rating system from 0 to 10, where 0 represents "no pain" and 10 represents the worst possible pain.

SECONDARY OUTCOMES:
The Zoster Brief Pain Inventory (ZBPI) | At baseline (before therapy), at 1 day of treatment,, at 7 days post-treatment, 30 days post-treatment, and 90 days post-treatment
  The Zoster Brief Pain Inventory (ZBPI) was used as the HZ-specific pain measure. The daily activity questionnaire included seven items: general activity, mood, walking ability, normal work, relationships with others, sleep, and enjoyment of life. Each question concerning daily activity was scored on a scale from 0 to 10, where 0 indicated no interference and 10 indicated complete interference.

CONTACTS AND LOCATIONS:
Locations (1):
- Inner Mongolia Baogang Hospital, Baotou, Inner Mongolia, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: January 2026-January 2031
Access Criteria: A proposal that describes planned analyses must be submitted or whether a data sharing agreement must be signed.

REFERENCES:
- [Background] Russo M, Graham B, Santarelli DM. Gabapentin-Friend or foe? Pain Pract. 2023 Jan;23(1):63-69. doi: 10.1111/papr.13165. Epub 2022 Oct 27. PMID 36300903
- [Background] Elhouty MG, Elbahrawy K, Elawady MS. Rhomboid intercostal block versus serratus block for postoperative analgesia after thoracoscopic sympathectomy for primary palmar hyperhidrosis: a randomized controlled trial. BMC Anesthesiol. 2023 Jul 19;23(1):241. doi: 10.1186/s12871-023-02203-z. PMID 37468840
- [Background] Rosamilia LL. Herpes Zoster Presentation, Management, and Prevention: A Modern Case-Based Review. Am J Clin Dermatol. 2020 Feb;21(1):97-107. doi: 10.1007/s40257-019-00483-1. PMID 31741185
- [Background] Asada H. Recent topics in the management of herpes zoster. J Dermatol. 2023 Mar;50(3):305-310. doi: 10.1111/1346-8138.16666. Epub 2022 Dec 20. PMID 36539935
- [Background] Okmen K, Gurbuz H, Ozkan H. Application of unilateral rhomboid intercostal and subserratus plane block for analgesia after laparoscopic cholecystectomy: a quasi-experimental study. Korean J Anesthesiol. 2022 Feb;75(1):79-85. doi: 10.4097/kja.21229. Epub 2021 Jul 20. PMID 34283910
- [Background] Wang X, Turner EL, Li F. Designing individually randomized group treatment trials with repeated outcome measurements using generalized estimating equations. Stat Med. 2024 Jan 30;43(2):358-378. doi: 10.1002/sim.9966. Epub 2023 Nov 27. PMID 38009329
- [Background] Patil A, Goldust M, Wollina U. Herpes zoster: A Review of Clinical Manifestations and Management. Viruses. 2022 Jan 19;14(2):192. doi: 10.3390/v14020192. PMID 35215786
- [Background] Li SJ, Feng D. Comparison of two distinct needle tip positions in pulsed radiofrequency for herpes zoster-related pain. CNS Neurosci Ther. 2023 Jul;29(7):1881-1888. doi: 10.1111/cns.14146. Epub 2023 Mar 7. PMID 36880287
- [Background] Boezaart AP, Lucas SD, Elliott CE. Paravertebral block: cervical, thoracic, lumbar, and sacral. Curr Opin Anaesthesiol. 2009 Oct;22(5):637-43. doi: 10.1097/ACO.0b013e32832f3277. PMID 19680122
- [Background] Xue M, Yuan R, Yang Y, Qin Z, Fu R. Application of ultrasound-guided thoracic paravertebral block or intercostal nerve block for acute herpes zoster and prevention of post-herpetic neuralgia: A case-control retrospective trial. Scand J Pain. 2024 Jul 9;24(1). doi: 10.1515/sjpain-2024-0030. eCollection 2024 Jan 1. PMID 38981512